CLINICAL TRIAL: NCT00226668
Title: A Phase III Randomized, Double-Blind Study Comparing Human Corticotropin-Releasing Factor (hCRF) to Dexamethasone for Control of Symptoms Associated With Peritumoral Brain Edema in Patients With Primary Malignant Glioma
Brief Title: XERECEPT® (hCRF) for Primary Glioma Patients Requiring Dexamethasone to Treat Peritumoral Brain Edema
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Alternate study projected to assess imaging endpoints versus clinical endpoints.
Sponsor: Celtic Pharma Development Services (Industry)
Collaborators: Neurobiological Technologies (Industry)
Responsible Party: Patrick Rossi, MD - Medical Monitor, Celtic Pharma Development Services
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTI 0302; corticorelin acetate injection
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2008-01-03 (Estimated); Status verified 2007-12

CONDITIONS: Brain Edema; Brain Tumor
Keywords: peritumoral brain edema; edema; malignant brain tumor; astrocytoma; brain tumor; dexamethasone; Decadron
MeSH Terms: conditions — Brain Edema; Brain Neoplasms; Edema; Astrocytoma | interventions — Corticotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Experimental): Patients will receive hCRf (XERECEPT) 2mg/day and dexamethasone 4 mg/day along with any open-label dexamethasone that they may be taking
  Interventions: Drug: hCRF
- II (Placebo Comparator): Patients will receive placebo hCRF (XERECEPT) 2mg/day and dexamethasone 4 mg/day along with any open-label dexamethasone they may be taking
  Interventions: Drug: placebo hCRF

INTERVENTIONS:
Drug: hCRF — hCRF 2mg/day; dexamethasone 4mg/day along with any open-label dexamethasone they may be taking
  Other Names: XERECEPT (corticorelin acetate injection)
  Arms: I
Drug: placebo hCRF — placebo hCRF 2mg/day, dexamethasone 4mg/day and any open-label dexamethasone they may be taking
  Other Names: placebo XERECEPT (corticorelin acetate injection)
  Arms: II

SUMMARY:
The purpose of this study is to examine the safety and efficacy of XERECEPT (human Corticotropin-Releasing Factor, or hCRF) compared to dexamethasone in patients with primary malignant glioma who require increased dexamethasone doses to control symptom of peritumoral brain edema.

DETAILED DESCRIPTION:
XERECEPT is not a potential treatment for cancer, but may reduce the edema associated with tumors and as a result, decrease neurological symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a primary malignant glioma.
* Symptomatic peritumoral brain edema requiring initiation or increase of dexamethasone treatment.
* If a patient is on dexamethasone for treatment of symptomatic peritumoral brain edema, the dose must be stable and should not exceed 24mg/dl for a minimum of 7 days prior to Baseline.
* Presence of peritumoral brain edema confirmed by MRI scan or comparable diagnostic technology obtained within 21 days of Baseline.
* Capable of self-administration of subcutaneous injections twice daily for 8 weeks or availability of assistance from caregiver.

Exclusion Criteria:

* Need for surgery, radiosurgery or radiation therapy or the introduction of new chemotherapeutic regime within 2 weeks of study treatment.
* Systemic steroid use for any other indication than peritumoral brain edema.
* Patients on dexamethasone or anticonvulsant therapy.
* Serious concomitant cardiovascular, pulmonary, renal, gastrointestinal or endocrine metabolic disease which could put the patient at unusual risk for study participation.
* Central nervous system (CNS) infection.
* Conditions that are considered contradictions for patients to receive niacin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-01; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the proportion of responders, i.e. patients in each treatment group who show improvement at the end of Week 1 and continue to be classified as improved relative to Baseline at Week 2. | Prospective

CONTACTS AND LOCATIONS:
Overall Officials: William Shapiro, MD, Principal Investigator — Barrow Neurological Institute
Locations (26):
- United States (24):
  - Barrow Neurological Institute, Phoenix, Arizona
  - UC San Diego Cancer Center, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University Medical Center, Palo Alto, California
  - UC Davis Medical Center, Sacramento, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Moffitt Cancer Center and Research, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Beth Israel Deaconess Med Center, Boston, Massachusetts
  - Field Neurosciences Institute, Saginaw, Michigan
  - Neurology Group of Bergen County, Ridgewood, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - Weill Medical College of Cornell University, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - University Hematology Oncology Care, LLC, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Clinic, Portland, Oregon
  - Methodist Healthcare - University Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Ottawa Regional Cancer Centre, Ottawa, Ontario